CLINICAL TRIAL: NCT00517452
Title: Phase 2-3 Observational Wound Care Study Comparing Application of Platelet Rich Plasma With Standard of Care Wound Closure in Vascular Patients Requiring a Groin Incision.
Brief Title: Platelet Rich Plasma Study in Lower Extremity Bypass Surgery
Acronym: PRP
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Dr. K. Lawlor, Lawson Health Research Institute
Other Study IDs: R-07-098
Record Dates: First submitted 2007-08-16; First posted 2007-08-17 (Estimated); Last update posted 2011-01-05 (Estimated); Status verified 2011-01

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Platelet Rich Plasma: Group received platelet rich plasma and observed over a period of 30 days or until wound closure
- Standard Wound Care: Group was treated as per standard care

SUMMARY:
The use of platelet rich plasma will decrease wound infection postop.

ELIGIBILITY:
Inclusion Criteria:

* Vascular surgical patients scheduled for elective lower extremity bypass surgery,aortoiliac revascularizations and endovascular AAA repair requiring a groin incision Exclusion Criteria:Patients requiring emergent procedures, unable to give informed consent

Ages: 35 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Vascular surgical patients scheduled for elective lower extremity bypass surgery,aortoiliac revascularizations and endovascular AAA repair requiring a groin incision
Sampling Method: Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2007-05; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Wound healing | 4- 6 weeks post op

CONTACTS AND LOCATIONS:
Overall Officials: Kirk D Lawlor, Principal Investigator — London Health Sciences Centre, University of Western Ontario